CLINICAL TRIAL: NCT00002377
Title: A Comparison of Valganciclovir and Ganciclovir in the Treatment of Cytomegalovirus (CMV) of the Eyes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: WV15376
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2005-07

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections | interventions — Valganciclovir; Ganciclovir

INTERVENTIONS:
Drug: Valganciclovir
Drug: Ganciclovir

SUMMARY:
To investigate the efficacy and safety of RS-79070 when used as induction therapy in patients with newly diagnosed peripheral retinitis. To assess the effects of induction and maintenance level dosing of RS-79070 on CMV viral load, estimated by plasma CMV PCR. To assess the pharmacokinetics of ganciclovir following administration of RS-79070 in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Documented AIDS diagnosis
* Newly diagnosed peripheral CMV retinitis
* More than 3 weeks of previous therapy for CMV retinitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-01 (Actual); Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (15):
  - Univ of California / Irvine, Irvine, California
  - Univ of California / San Diego / Dept of Pediatrics, La Jolla, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Davies Med Ctr / Institute for HIV Research, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - QUEST Clinical Research, San Francisco, California
  - Dr Alan Palestine, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Eye Clinic, Atlanta, Georgia
  - New England Med Ctr, Boston, Massachusetts
  - New York Univ Med Ctr, New York, New York
  - St Luke's - Roosevelt Hosp Ctr / Div of Infect Dis, New York, New York
  - New York Hosp - Cornell Med Ctr, New York, New York
  - Duke Univ Eye Ctr, Durham, North Carolina
  - Austin Infectious Disease Consultants, Austin, Texas
- Canada (4):
  - St Pauls Hosp, Vancouver, British Columbia
  - The Toronto Hosp / Dept of Infectious Disease, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec
  - Royal Victoria Hosp, Montreal, Quebec